CLINICAL TRIAL: NCT07370103
Title: Carotid Artery Corrected Flow Time and Respiratory Variation of Blood Flow Peak Velocity for Prediction of Hypotension After Induction of General Anaesthesia in Adult Patients With Chronic Liver Disease
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ismail Mohammed, assisstant proffesor of anaesthesia, Ain Shams University
Other Study IDs: FMASU R331/2025; ain shams university (Registry Identifier: ain shams university)
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hypotension on Induction
Keywords: carotid time,respiratory variation,hypotension,chronic liver disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients presented with hypotension after induction of general anaesthesia: POST INDUCTION HYPOTENSION (PIH ) group
- patients not presented by hypotension after induction of general anaesthesia: NON POST INDUCTION HYPOTENSION (NON PIH GROUP)

SUMMARY:
Baseline Measurements

For the ultrasound parameters, it is the average of three readings In supine position .

The investigators will continuously monitoring during induction and 10 minutes after.

Hemodynamic Monitoring:

* Heart rate from ECG
* SpO2
* Etco2
* Blood pressure . invasive Blood pressure
* The radial artery level is the site of continuous arterial pressure monitoring with an arterial catheter.
* Ultrasound Measurements:

The patient will be positioned in a supine position, with the right side of the neck completely exposed. The transverse part Of the main carotid artery beneath the thyroid cartilage will be precisely identified using ultrasound device (sonosite edge portablp.fojy usa)via a linear array probe (4-15 MHz), with the marker directed toward the patient's head. Thus, the sampling line will be positioned at the center of the carotid lumen, around 2 cm from the carotid bifurcation, and the electronic angle correction cursor will be pointed in the direction of blood flow. Insonation angles between the ultrasound beam and blood flow will be maintained at or < 60°. Next, the carotid blood flow waveform will be acquired, and the consecutive stable carotid pulse Doppler flow spectrum will be determined with an optimal level of image quality.

The Correction: To get the corrected carotid flow time (ccFT), the measured FT will be adjusted for the patient's heart rate (HR). A commonly used formula is Wodey's formula.

A single, experienced sonographer will perform all measurements, and a subset of measurements will be reviewed by a second blinded observer to assess inter-rater reliability."

Peak Velocity: Measure the peak systolic blood flow velocity at the same location.

Respiratory Variation (ΔVpeak): Calculate the difference between the maximum and minimum peak velocities during a single respiratory cycle: \Delta V_{peak} = (V_{peak(max)} - V_{peak(min)}) / ((V_{peak(max)} + V_{peak(min)})/2) \times 100\%. The patient should be asked to breathe normally during this measurement.

Flow time (FT), which is known as the time period between the systolic increase phase and dicrotic notch, was calculated and then adjusted for heart rate (HR) via equations outlined below.

Wodey's (W) equation∶ FTc(W) = FT + 1.29 ∗ (HR - 60)

Anasthesia:

Patients will have routine fasting for at least 6 to 8 h and will not allowed to drink any solution or fluid 2 to 4 h prior to surgery.

No premedication will be given A standardized induction protocol will be used. At the operating theatre, a three-lead electrocardiogram (ECG), pulse oximetry (SpO2), and noninvasive arterial pressure monitoring will be applied.

After pre-oxygenation for 5 min anesthesia induction of propofol 1_2mg , fentanyl 1 ug/kg, and 0.15 mg/kg cisatracurium . After 3 min of mask ventilation, direct laryngoscopy will be employed for tracheal intubation. . Respiratory setting of anesthesia machine (Aestiva, GE/Datex-Ohmeda) will be set as follows: volume-controlled ventilation (VCV), inspiratory-expiratory (I:E) ratio of 1:2, respiratory rate of 8-10 bpm, tidal volume of 8 mL/kg of ideal weight [45.5 + 0.91x (height in cm-152.4)], and PEEP of 5 cm H2O in 50% oxygen with air. Respiratory settings will be adjusted to maintain the PETCO2 at less than 50 mmHg. Anesthesia will be maintained with sevoflurane (1.5-2.5%) and intermittent injection of cisatracurium 0.02mg/kg as needed to keep the entropy scale between 40 and 60 and for muscle relaxation. The mean arterial pressure was kept between 60 and 80 mmHg.

Hemodynamic Data Collection: Invasive mean arterial pressure (MAP) will be continuously recorded for 5-10 minutes post-induction.

Hypotension Definition: Hypotension will be defined as a decrease in MAP by >20% from the baseline value or an absolute MAP of <65 mmHg for more than one minute.This definition is clinically relevant and widely used in the anesthesia literature.

Postinduction hypotension will be treated with 250 ml saline iv boluse repeated if successfully restore blood pressure.

If refractory to fluid we will inject intravenous ephedrine in 3 mg bolus doses and repeated when necessary.

Significant bradycardia (heart rate < 40 beats/min) will be treated with intravenous boluses of atropine (0.5 mg).

Study duration 3 months or end of recruitment of sample

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients (≥ 18 years) with a confirmed diagnosis of CLD (e.g., cirrhosis, non-alcoholic steatohepatitis)

  * scheduled for elective surgery under general anesthesia.
  * ASA 2,3,4
  * ASA 4 patients will be included only if their baseline MAP is >65 mmHg, as per the exclusion criteria

Exclusion Criteria:

* • Refusal to participate

  * Patients with known cardiac disease (e.g., severe valvular disease, congestive heart failure),
  * pre-existing severe hypotension (e.g., mean arterial pressure <65 mmHg
  * emergency surgery
  * anatomical variations preventing adequate ultrasound visualization of the carotid artery.
  * Carotid artery stenosis.
  * Mean arterial pressure (MAP) > 120 mmHg before anesthesia
  * any previous record of neck surgery or trauma.
  * acute renal injury.
  * oral angiotensin receptor blockers or angiotensin-converting enzyme inhibitors (ACEI)
  * lateral, prone, and lithotomy operations
  * body mass index (BMI) > 30 kg/m2 or < 15 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Adult patients (≥ 18 years) with a confirmed diagnosis of CLD (e.g., cirrhosis, non-alcoholic steatohepatitis)
  * scheduled for elective surgery under general anesthesia.
  * ASA 2,3,4
  * ASA 4 patients will be included only if their baseline MAP is >65 mmHg, as per the exclusion criteria
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
prediction of hypotension | 3 months
  Prediction of hypotension after induction of anesthesia by receiver operating characteristic curves of the carotid artery FTc and ΔVpeak Logistic regression analysis Cutoff value for liver disease patients

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No